| Exploring the Role of a Second-Generation Mindfulness-Based Intervention for Improving Quality of Life, Pain Management, and Psycho-Spiritual Wellbeing in Cancer Patients: A Mixed-Methods investigation |
|---|
| Document date: 01/11/2024 |

## **Consent Form**

**Study Title:** Exploring the Role of a Second-Generation Mindfulness-Based Intervention for Improving Quality of Life, Pain Management, and Psycho-Spiritual Wellbeing in Cancer Patients: A Mixed-Methods Investigation

In order to complete the consent form below, please create a unique ID code.

This will be comprised of the first two letters of your first name and the last three digits of your telephone number. For example, if your first name was Roy and your phone number 07630 435 925, your unique 5-digit code would be RO925.

| Participant Unique Code: |
|---|
| Participant Name: |
| Participant Consent: □ |
| Date: |
| Participant telephone number: |
| I confirm that I have read and understood the participant information sheet for the above study. I have had the opportunity to ask questions, and all my questions have been answered satisfactorily. |
| □ I confirm |
| I understand that my participation in this study is voluntary and that I am free to withdraw at any time without giving any reason, up until two weeks after my participation, without any adverse effects. |
| □ I confirm |
| I understand the protocol of a Randomised Controlled Trial and understand that I will not know which intervention group I am in/ have been in until the end of the intervention period. |
| I agree to take part in the Meditation Awareness Training (MAT) program if assigned to the intervention group, or to be placed into a treatment as usual group if assigned to the control group, understanding that I will have the opportunity to participate in the MAT program after the study period. |
| □ I confirm |

| I understand that this study involves completing online questionnaires at several time points and may involve submitting an online diary and participating in telephone interviews to discuss my experiences. |
|---|
| □ I confirm |
| I consent to the use of my anonymized data for research purposes, including publications and presentations related to this study. |
| □ I confirm |
| I understand that all information I provide will be kept confidential and stored securely. Only the research team will have access to my data, and it will be used only for the purpose of this study. |
| I understand that the results of the study will be published in a way that I cannot be identified. |
| I agree that my anonymized data may be used for future research by this research team. |
| I understand that upon the completion of the study I will be invited and may enter into a prize draw to win a £50 shopping voucher, which be drawn at random. $\Box$ I confirm |
| For further information or to withdraw from the study, I understand that I can contact: |
| Researcher: Chloe Wells |
| Email: chloe.wells2@derby.ac.uk |
| Supervisor: Dr William Van Gordon |
| Email: W.VanGordon@derby.ac.uk |
| Telephone: +44 (0)1332 591066 |

Thank you for your participation in this study.